CLINICAL TRIAL: NCT01133860
Title: An Exploratory Phase II Dose Escalation Study of Eltrombopag in MYH9 Related Disease
Brief Title: Efficacy of Eltrombopag to Improve Thrombocytopenia of MYH9-related Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Pavia (Other); GlaxoSmithKline (Industry); Azienda Ospedaliera di Padova (Other); Azienda Ospedaliera di Perugia (Other); Fondazione Telethon (Other)
Responsible Party: Prof. Carlo Balduini, Head of the Unit of Internal Medicine III, IRCCS Policlinico San Matteo Foundation, Pavia, Italy, IRCCS Policlinico San Matteo Foundation, Pavia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eltrombopag-MYH9-2008
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Blood Platelet Disorders
Keywords: inherited thrombocytopenia; MYH9 mutations; eltrombopag
MeSH Terms: conditions — Blood Platelet Disorders | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eltrombopag (Experimental)
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — Eltrombopag, administered orally, 50 mg/daily for 21 days. Patients with platelet counts between 100 and 150x10e9/L at day 21 will continue eltrombopag 50 mg/daily for 21 additional days. Patients with platelet count lower than 100x10e9/L at day 21 will receive eltrombopag 75 mg/daily for additional 21 days. Patients with more than 150x10e9 platelets/L at day 21 will stop therapy.
  Other Names: Revolade; Promacta

SUMMARY:
The term MYH9-related disease (MYH9RD) includes four genetic disorders: May-Hegglin anomaly, Sebastian syndrome, Fechtner syndrome, and Epstein syndrome. All these disorders derive from mutation of a unique gene, named MYH9, and they have been recognized as different clinical presentations of a single illness that was named MYH9RD. All patients affected by MYH9RD present since birth with thrombocytopenia, which can result in a variable degree of bleeding diathesis; some of them subsequently develop additional clinical manifestations, such as renal damage, sensorineural hearing loss, and/or presenile cataracts. Eltrombopag is an oral thrombopoietin receptor agonist that stimulates proliferation and differentiation of megakaryocytes, the bone marrow cells that produce blood platelets. This drug is effective in increasing platelet count in healthy volunteers, as well as in patients affected by some acquired thrombocytopenias, such as idiopathic thrombocytopenic purpura and HCV related thrombocytopenia. The purpose of this study is to determine if eltrombopag, administered orally at the dose of 50 or 75 mg/daily for up to 6 weeks, is effective in increasing platelet count of patients affected by MYH9RD. Further aims of this study are to test if eltrombopag is effective in reducing bleeding tendency of MYH9RD patients; to evaluate safety and tolerability of eltrombopag in patients with MYH9RD; to evaluate in vitro function of platelets produced during therapy in patients responding to this drug.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or more
* Confirmed diagnosis of MYH9-related disease
* Average platelet count for the previous year less than 50x10e9/L
* Written informed consent

Exclusion Criteria:

* Diseases known to involve the risk of thromboembolic events (e.g. atrial fibrillation)
* History of thrombosis within 1 year
* Use of drugs that affect platelet function (including but not limited to, aspirin, clopidogrel or NSAIDS) or anti-coagulants
* Females who are pregnant or nursing (a negative pregnancy test in required before enrollment of fertile women)
* Formal refusal of any recommendation of a safe contraception
* Alcohol or drug addiction
* Altered renal function as defined by creatinine of 20 mg/L or more
* Any other disease or condition that by the advise of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for the study, including physical, psychiatric, social and behavioral problems. HCV positivity and liver diseases will not be considered an exclusion criterion since a phase II study showed that eltrombopag was effective and safe in this patient population.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Balduini, MD, Principal Investigator — IRCCS Policlinico San Matteo Foundation, Pavia, Italy
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Padova, Unità di Medicina Generale e Patologia Speciale, Padua
  - Fondazione IRCCS Policlinico San Matteo, Unità di Medicina III, Pavia
  - Policlinico Monteluce, Sezione di Medicina Interna e Cardiovascolare, Perugia

REFERENCES:
- [Background] Seri M, Cusano R, Gangarossa S, Caridi G, Bordo D, Lo Nigro C, Ghiggeri GM, Ravazzolo R, Savino M, Del Vecchio M, d'Apolito M, Iolascon A, Zelante LL, Savoia A, Balduini CL, Noris P, Magrini U, Belletti S, Heath KE, Babcock M, Glucksman MJ, Aliprandis E, Bizzaro N, Desnick RJ, Martignetti JA. Mutations in MYH9 result in the May-Hegglin anomaly, and Fechtner and Sebastian syndromes. The May-Heggllin/Fechtner Syndrome Consortium. Nat Genet. 2000 Sep;26(1):103-5. doi: 10.1038/79063. PMID 10973259
- [Background] Seri M, Savino M, Bordo D, Cusano R, Rocca B, Meloni I, Di Bari F, Koivisto PA, Bolognesi M, Ghiggeri GM, Landolfi R, Balduini CL, Zelante L, Ravazzolo R, Renieri A, Savoia A. Epstein syndrome: another renal disorder with mutations in the nonmuscle myosin heavy chain 9 gene. Hum Genet. 2002 Feb;110(2):182-6. doi: 10.1007/s00439-001-0659-1. Epub 2001 Dec 14. PMID 11935325
- [Background] Seri M, Pecci A, Di Bari F, Cusano R, Savino M, Panza E, Nigro A, Noris P, Gangarossa S, Rocca B, Gresele P, Bizzaro N, Malatesta P, Koivisto PA, Longo I, Musso R, Pecoraro C, Iolascon A, Magrini U, Rodriguez Soriano J, Renieri A, Ghiggeri GM, Ravazzolo R, Balduini CL, Savoia A. MYH9-related disease: May-Hegglin anomaly, Sebastian syndrome, Fechtner syndrome, and Epstein syndrome are not distinct entities but represent a variable expression of a single illness. Medicine (Baltimore). 2003 May;82(3):203-15. doi: 10.1097/01.md.0000076006.64510.5c. PMID 12792306
- [Background] Bussel JB, Cheng G, Saleh MN, Psaila B, Kovaleva L, Meddeb B, Kloczko J, Hassani H, Mayer B, Stone NL, Arning M, Provan D, Jenkins JM. Eltrombopag for the treatment of chronic idiopathic thrombocytopenic purpura. N Engl J Med. 2007 Nov 29;357(22):2237-47. doi: 10.1056/NEJMoa073275. PMID 18046028
- [Background] McHutchison JG, Dusheiko G, Shiffman ML, Rodriguez-Torres M, Sigal S, Bourliere M, Berg T, Gordon SC, Campbell FM, Theodore D, Blackman N, Jenkins J, Afdhal NH; TPL102357 Study Group. Eltrombopag for thrombocytopenia in patients with cirrhosis associated with hepatitis C. N Engl J Med. 2007 Nov 29;357(22):2227-36. doi: 10.1056/NEJMoa073255. PMID 18046027
- [Derived] Pecci A, Gresele P, Klersy C, Savoia A, Noris P, Fierro T, Bozzi V, Mezzasoma AM, Melazzini F, Balduini CL. Eltrombopag for the treatment of the inherited thrombocytopenia deriving from MYH9 mutations. Blood. 2010 Dec 23;116(26):5832-7. doi: 10.1182/blood-2010-08-304725. Epub 2010 Sep 15. PMID 20844233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled between January 2009 and January 2010 as outpatients in medical clinic
Groups:
- Eltrombopag: Eltrombopag, administered orally, 50 mg/daily for 21 days. Patients with platelet counts between 100 and 150x10e9/L at day 21 continued eltrombopag 50 mg/daily for 21 additional days. Patients with platelet count lower than 100x10e9/L at day 21 received eltrombopag 75 mg/daily for additional 21 days. Patients with more than 150x10e9 platelets/L at day 21 stopped therapy.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.0 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  Italy | 12

OUTCOME MEASURES:

1. Primary Outcome: Response to Drug Based on Platelet Count at the End of Therapy
Description: The primary endpoints were the achievement of a platelet count over 100 x10e9/L or at least 3 times the baseline value (major response), or at least twice the baseline value but less than major response (minor response). The overall response to therapy is reported. Platelet count was measured at the end of therapy (21 or 42 days, see study design) by phase-contrast microscopy.
Time Frame: 21 days and/or 42 days of therapy, 15 and 30 days after the end of therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
percentage of participants | 91.6 [61.5 to 99.7]

2. Secondary Outcome: Bleeding Tendency Assessed by WHO Bleeding Score
Description: The percentage of patients with bleeding diathesis (grade 1, i.e. cutaneous bleeding, or grade 2, i.e. mild blood loss, according to WHO bleeding score) was calculated at baseline and at the end of therapy. The results are expressed as the mean change in the percentage of patients with bleeding diathesis (95%CI).
Time Frame: 21 days and/or 42 days of therapy, 15 and 30 days after the end of therapy
Measure: Mean (95% Confidence Interval); unit: participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
participants | 66.7 [31.7 to 100]

3. Secondary Outcome: All Types of Adverse Events
Description: All type of adverse events were registered.Results indicate the number of participants who experience a side effect of the drug.
Time Frame: 21 days and/or 42 days of therapy, 15 and 30 days after the end of therapy
Measure: Number; unit: number of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
number of participants | 2

4. Secondary Outcome: in Vitro Function of Platelets Produced During Therapy in Responding Patients
Description: in vitro platelet function will be assessed in patients achieving a platelet count of 100 x10e9/L or more at the end of the therapy
Time Frame: 21 days or 42 days of therapy
Measure: Number; unit: participants
Groups:
- Eltrombopag: In patients with more than 100 x10e9 platelets/L at the end of therapy, we evaluated also the in vitro platelet aggregation after stimulation with adenosine diphosphate (5 and 20 mcM), collagen (5 and 20 mg/mL) and ristocetin (3 mg/mL) by the densitometric method of Born in native platelet rich plasma. The extent of platelet aggregation was measured 5 minutes after the addition of stimulating agents and results obtained in patients were compared with the normal ranges in the laboratories where the assay was performed. Results are reported as the number of patients with normal platelet aggregation.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 7
participants | 5

ADVERSE EVENTS:
Time Frame: 51 or 72 days, i.e. during the administration of Eltrombopag (21 or 42 days, see study design) and until 30 days after the end of treatment (see study design).
Arm/Group | Eltrombopag
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=12)
headache (General disorders) | 2 (2) — mild and transient headache at the beginning of the treatment, duration 3-4 days, spontaneous remission
dry mouth (General disorders) | 1 (1) — transient sensation o dry mouth at the beginning of the treatment, duration 3-4 days, spontaneous remission

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes